CLINICAL TRIAL: NCT05060614
Title: MOLECULAR BIOMARKERS IN DELIRIUM AND DEMENTIA
Brief Title: Analyses of Cerebrospinalfluid in Patients With Delirium
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Leiv Otto Watne, Postdoctoral Research Fellow, Oslo University Hospital
Other Study IDs: 2016/1368
Record Dates: First submitted 2021-06-30; First posted 2021-09-29 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CSF, blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Hip fracture surgery — Hip fracture surgery

SUMMARY:
The current project aims to measure biomarkers in the cerebrospinalfluid (CSF) and serum samples from patients with delirium. We hope to uncover new insights into the pathophysiology of delirium and explore its link to dementia.

DETAILED DESCRIPTION:
Delirium is a common and serious complication to acute illness, and is characterized by acute disturbances in attention, awareness, and cognition. Dementia is a major risk factor of delirium, and delirium increases the risk of dementia progression and development. As the conditions share both clinical and epidemiological features, some researchers suggest that also pathophysiological links are shared. Understanding delirium pathophysiology, which is poorly understood, may thus help elucidate early molecular mechanisms in dementia.

This study aims to to increase our understanding of the pathophysiology of delirium and molecular links between delirium and dementia, by exploring cerebrospinal fluid (CSF) biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute hip fracture

Exclusion Criteria:

* Moribund patients.
* Lack of consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients acutely admitted with a hip fracture.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Delirium | Daily during hospital stay (pre-/and postoperatively) until 5 days after surgery (or discharge)
  Pre- and postoperative delirium

SECONDARY OUTCOMES:
Dementia | Cognitive changes the first 48 months after inclusion
  Incident dementia

CONTACTS AND LOCATIONS:
Overall Officials: Leiv O Watne, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Leiv Otto Watne, Oslo, Other, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Availability is dependent on approval from the Regional Committee for Medical and Health Research Ethics in Norway. The data are not publicly available due to privacy or ethical restrictions.